CLINICAL TRIAL: NCT03389750
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Crossover Study to Evaluate the Abuse Potential of Oxymorphone Compared to Other Mu Opioid Agonists in Physically Dependent Opioid Users With Moderate-to-Severe Opioid Use Disorder
Brief Title: A Study to Evaluate the Abuse Potential of Oxymorphone Compared to Other Mu Opioid Agonists.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Sandra D. Comer, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 7565
Record Dates: First submitted 2017-12-19; First posted 2018-01-04 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxycodone; Oxymorphone; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Intravenous Challenge Drug
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intravenous Challenge Drug: Oxymorphone (Active Comparator): Intravenous (IV) Dose Range: 1.8, 3.2, 5.6, 10 mg/70kg of the participant's body weight
  Interventions: Drug: Intravenous Challenge Drug
- Intravenous Challenge Drug: Oxycodone (Active Comparator): IV Dose Range: 10, 18, 32, 56 mg/70kg of the participant's body weight
  Interventions: Drug: Intravenous Challenge Drug
- Intravenous Challenge Drug: Hydromorphone (Active Comparator): IV Dose Range: 3.2, 5.6, 10, 18 mg/70kg of the participant's body weight
  Interventions: Drug: Intravenous Challenge Drug
- Intravenous Challenge Drug: Placebo (Placebo Comparator): IV saline
  Interventions: Drug: Intravenous Challenge Drug

INTERVENTIONS:
Drug: Intravenous Challenge Drug — Intravenous administration of opioid drugs (oxycodone, oxymorphone, hydromorphone), for the purpose of comparison of their abuse potential among each other, and in comparison to placebo (saline).
  Other Names: Oxycodone, Oxymorphone, Hydromorphone, or Placebo

SUMMARY:
Significant public health concerns have arisen from the intravenous misuse of oxymorphone, a potent mu-opioid pain medication. However, little is known about its abuse potential relative to other mu-opioid analgesics. The present study is designed to examine the abuse liability of intravenous oxymorphone compared to other mu opioid agonists (oxycodone, and hydromorphone) among physically dependent opioid abusers.

DETAILED DESCRIPTION:
Significant public health concerns have arisen from the misuse of oxymorphone, a potent mu-opioid pain medication approved by the Food and Drug Administration as Opana and Opana ER. However, little is known about its abuse potential relative to other mu opioid analgesics. The present study is designed to examine the abuse liability of intravenous oxymorphone compared to other mu opioid agonists (oxycodone and hydromorphone). Participants who are physically dependent on opioids and who meet DSM 5 criteria for Opioid Use Disorder will complete the study across 2 sites, New York State Psychiatric Institute (NYSPI) and the University of Kentucky; a total of 6 additional participants across 2 sites will complete a pilot phase of the study in order to establish comparable opioid dose-response functions based on subjective ratings of Drug Liking. All participants will reside in clinical inpatient units for the duration of the studies (both the 8- to 9-week main and 4- to 5-week pilot studies; please note that the pilot study is identical in design to the first 4-5 weeks of the main study). The study design is based on the 2017 FDA Assessment of Abuse Potential of Drugs: Guidance for Industry [Center for Drug Evaluation and Research (CDER), 2017], which suggests the use of a double-blind, positive- and placebo-controlled design that includes a qualification phase and VAS measure of Drug Liking. The proposed study also examines the reinforcing effects of oxymorphone and other mu opioid agonists using two different drug self-administration procedures, namely Drug versus Money and Drug versus Drug choice procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide signed and dated written consent.
2. Self-reported opioid use for nontherapeutic purposes on at least 21 days in the 30 days prior to screening, physical dependence on opioids, recent intravenous opioid use, and meeting DSM 5 criteria for moderate-severe opioid use disorder.
3. Positive urine drug screen for opioids (those who are in a methadone or buprenorphine treatment program are ineligible; physical dependence on street methadone or buprenorphine are also exclusionary so participants must produce at least one methadone- or buprenorphine-negative urine during screening).
4. ≥ 21 and ≤ 55 years of age.
5. Body mass index (BMI) ≥ 18 and ≤ 35 kg/m2 and weight ≥ 50 kg (110 pounds).
6. Otherwise healthy as determined by the investigator.
7. Demonstrate understanding how to complete the self-administration tasks and VAS Questionnaire.
8. Women of childbearing potential must not be pregnant or breastfeeding at screening.
9. Willing and able to comply with all testing requirements defined in the protocol.

participation in the Study Treatment Phase:

1. During the Study Qualification Phase, on the bipolar 100--mm Drug Liking VAS, the subject must provide Emax ≥ 40 mm and < 60 mm following placebo and, following morphine 56 mg/70 kg, i.v., Emax ≥ 60 mm and ≥ 15 mm closer to "Strong Liking" than the Emax to placebo.
2. In the judgment of the investigator, the subject is able to tolerate the i.v., opioids administered in the study, including the ability to complete most pharmacodynamics assessments administered post--dose.
3. In the judgment of the study staff, the subject's general behavior during the Study Qualification Phase suggests the ability to successfully complete the Study Treatment Phase.

Exclusion Criteria:

1. History of a medical or psychiatric disorder that would prevent successful completion of the study.
2. Current DSM-5 diagnosis of substance use disorders requiring medical management other than OUD.
3. Suicidal ideation or intent with or without a plan at Screening or within 6 months prior to Screening (i.e., answering "Yes" to questions 4 and/or 5 on the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale).
4. Currently seeking or participating in treatment for substance use disorder.
5. Physically dependent on drugs of abuse (other than opioids, nicotine, or caffeine) or alcohol.
6. Medically important deviation from normal limits on physical examination, vital signs, screening laboratory tests, or 12--lead ECG.
7. Significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, or neurologic disorder.
8. Any surgical, or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test drug.
9. Family history of long QT syndrome and/or unexpected sudden cardiac death or is known to have QTc > 500 ms at screening.
10. Used an investigational agent within 30 days or 5 therapeutic half-lives of that agent, whichever is longer, prior to the first dose of study drug.
11. Hypersensitivity to opioids or any drug intended for use in this study.
12. Acute gastrointestinal symptoms (e.g., nausea, vomiting, fever, or Diarrhea unrelated to opioid withdrawal) ≤ 7 days before Day 1.
13. Any of the following values for laboratory tests at Screening:

    1. A positive pregnancy test in women of childbearing potential.
    2. Hemoglobin < 11 g/dL in males and < 10 gm/dL in females.
    3. Neutrophil count < 1.0 × 109/L.
    4. Platelet count < 75 × 109/L.
    5. Creatinine clearance < 50 ml/min per modified Cockcroft-Gault equation.
    6. Aspartate aminotransferase or alanine aminotransferase > 3.0x upper limit of normal.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — New York State Psychiatric Institute / Columbia University Medical Center
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - New York State Psychiatric Institute in the Division on Substance Use Disorders, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This investigation was a within-subjects design. The participants were presented with the following drugs/doses in randomized order: Oxymorphone (1.8, 3.2, 5.6, and 10 mg/70 kg) Oxycodone (10, 18, 32, 56 mg/70 kg) Hydromorphone (3.2, 5.6, 10, and 18 mg/70 kg) Placebo (0 mg). Data are only presented for individuals who received all 13 dose conditions (i.e., N=8).
Groups:
- Intravenous Challenge Drug: Oxycodone, oxymorphone, hydromorphone and placebo were administered in random order. A morphine condition was dropped prior to the initiation of the trial.
Period: Overall Study
Arm/Group | Intravenous Challenge Drug
Started | 16
Oxycodone | 8
Oxymorphone | 8
Hydromorphone | 8
Placebo | 8
Completed | 8
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Baseline demographics include all participants who were randomized/enrolled.
Groups:
- Intravenous Challenge Drug: All participants received: oxycodone, oxymorphone, and hydromorphone for the purpose of comparison of their abuse potential among each other and to placebo (saline).
Arm/Group | Intravenous Challenge Drug
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Positive Subjective Drug Effects (i.e., Drug "Liking").
Description: The positive subjective effects of the most efficacious dose of the intravenous challenge drugs. These are measured using self-reported assessment by the participant in terms of drug "liking" rated on a visual analog scale of 0-100. Higher values indicate a greater drug effect.
Time Frame: Throughout study enrollment period (8-9 weeks)
Population: The most robust self-reported drug "Liking" across the various dose of each IV drug (Scale: 0-100). These data are reported only for study completers (i.e., those individuals who experienced all 13 drug & dose drug conditions). Higher values indicate a greater drug effect.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- IV Placebo: Intravenous administration of placebo (saline, 0 mg/70kg)
- IV Oxymorphone 1.8 mg: Intravenous administration of Oxymorphone 1.8 mg/70kg.
- IV Oxymorphone 3.2 mg: Intravenous administration of Oxymorphone 3.2 mg/70kg.
- IV Oxymorphone 5.6 mg: Intravenous administration of Oxymorphone 5.6 mg/70kg.
- IV Oxymorphone 10 mg: Intravenous administration of Oxymorphone 10 mg/70kg.
- IV Hydromorphone 3.2 mg: Intravenous administration of Hydromorphone 3.2 mg/70kg.
- IV Hydromorphone 5.6 mg: Intravenous administration of Hydromorphone 5.6 mg/70kg.
- IV Hydromorphone 10 mg: Intravenous administration of Hydromorphone 10 mg/70kg.
- IV Hydromorphone 18 mg: Intravenous administration of Hydromorphone 18 mg/70kg.
- IV Oxycodone 10 mg: Intravenous administration of Oxycodone 10 mg/70kg.
- IV Oxycodone 18 mg: Intravenous administration of Oxycodone 18 mg/70kg.
- IV Oxycodone 32 mg: Intravenous administration of Oxycodone 32 mg/70kg.
- IV Oxycodone 56 mg: Intravenous administration of Oxycodone 56 mg/70kg.
Arm/Group | IV Placebo | IV Oxymorphone 1.8 mg | IV Oxymorphone 3.2 mg | IV Oxymorphone 5.6 mg | IV Oxymorphone 10 mg | IV Hydromorphone 3.2 mg | IV Hydromorphone 5.6 mg | IV Hydromorphone 10 mg | IV Hydromorphone 18 mg | IV Oxycodone 10 mg | IV Oxycodone 18 mg | IV Oxycodone 32 mg | IV Oxycodone 56 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
units on a scale | 52.1 (1.0) | 57.5 (2.8) | 71.8 (5.2) | 71.5 (6.1) | 84 (4.9) | 66.3 (3.8) | 71.3 (4.9) | 84.3 (4.8) | 79.6 (5.4) | 59.5 (3.9) | 63.3 (3.9) | 70.3 (4.4) | 79.1 (5.5)
Statistical Analysis 1: Comparison: IV Placebo vs IV Oxymorphone 1.8 mg vs IV Oxymorphone 3.2 mg vs IV Oxymorphone 5.6 mg vs IV Oxymorphone 10 mg vs IV Hydromorphone 3.2 mg vs IV Hydromorphone 5.6 mg vs IV Hydromorphone 10 mg vs IV Hydromorphone 18 mg vs IV Oxycodone 10 mg vs IV Oxycodone 18 mg vs IV Oxycodone 32 mg vs IV Oxycodone 56 mg; Test type: Equivalence — An F-test was used to assess for significant differences among the 13 dose conditions; p = .0001, ANOVA; F = 7.06 (DF=12)

ADVERSE EVENTS:
Time Frame: Throughout the 8-week inpatient period.
Groups:
- IV Challenge Drug: Placebo 0 mg: Intravenously administered saline solution.
- IV Challenge Drug: Oxymorphone 1.8 mg: Intravenously administered oxymorphone 1.8 mg/70kg
- IV Challenge Drug: Oxymorphone 3.2 mg: Intravenously administered oxymorphone 3.2 mg/70kg
- IV Challenge Drug: Oxymorphone 5.6 mg: Intravenously administered oxymorphone 5.6 mg/70kg
- IV Challenge Drug: Oxymorphone 10 mg: Intravenously administered oxymorphone 10 mg/70kg
- IV Challenge Drug: Hydromorphone 3.2 mg: Intravenously administered Hydromorphone 3.2 mg/70 mg/70kg
- IV Challenge Drug: Hydromorphone 5.6 mg: Intravenously administered Hydromorphone 5.6 mg/70 mg/70kg
- IV Challenge Drug: Hydromorphone 10 mg: Intravenously administered Hydromorphone 10 mg/70
- IV Challenge Drug: Hydromorphone 18 mg: Intravenously administered Hydromorphone 18 mg/70
- IV Challenge Drug: Oxycodone 10 mg: Intravenously administered oxycodone 10 mg/70 kg
- IV Challenge Drug: Oxycodone 18 mg: Intravenously administered oxycodone 18 mg/70 kg
- IV Challenge Drug: Oxycodone 32 mg: Intravenously administered oxycodone 32 mg/70 kg
- IV Challenge Drug: Oxycodone 56 mg: Intravenously administered oxycodone 56 mg/70 kg
Arm/Group | IV Challenge Drug: Placebo 0 mg | IV Challenge Drug: Oxymorphone 1.8 mg | IV Challenge Drug: Oxymorphone 3.2 mg | IV Challenge Drug: Oxymorphone 5.6 mg | IV Challenge Drug: Oxymorphone 10 mg | IV Challenge Drug: Hydromorphone 3.2 mg | IV Challenge Drug: Hydromorphone 5.6 mg | IV Challenge Drug: Hydromorphone 10 mg | IV Challenge Drug: Hydromorphone 18 mg | IV Challenge Drug: Oxycodone 10 mg | IV Challenge Drug: Oxycodone 18 mg | IV Challenge Drug: Oxycodone 32 mg | IV Challenge Drug: Oxycodone 56 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT03389750/Prot_SAP_000.pdf